CLINICAL TRIAL: NCT01486927
Title: A Phase I/III Open-label, Multicenter, Crossover Safety, Efficacy and Pharmacokinetic Study of Recombinant Coagulation Factor VIII (rFVIII) Compared to Recombinant Human Antihaemophilic Factor VIII (rFVIII; INN: Octocog Alfa) in Subjects With Hemophilia A, and a Repeat PK, Safety and Efficacy Study
Brief Title: An Open-label Safety, Efficacy and Pharmacokinetic Study of a Recombinant FVIII Compared to Recombinant Human Antihemophilic FVIII in Patients With Severe Hemophilia A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL627_1001; 2011-002393-23 (EudraCT Number)
Record Dates: First submitted 2011-11-19; First posted 2011-12-07 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-06

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; DNA, Ribosomal

ARMS (1):
- Recombinant Factor VIII (rFVIII) (Experimental)
  Interventions: Biological: rVIII-SingleChain; Biological: Octocog alfa

INTERVENTIONS:
Biological: rVIII-SingleChain — In Part 1 of the study, subjects received a single intravenous infusion of 50 IU/kg recombinant, single-chain coagulation factor VIII (rVIII-SingleChain) preceded by a 4-day washout period. In Parts 2 and 3 of the study, subjects received repeat injections of rVIII-SingleChain either as an on-demand or prophylaxis regimen at a dose and frequency determined by their study doctor. Subjects participating in the Part 3 PK analyses received a single infusion of 50 IU/kg rVIII-SingleChain and a repeat dose of the same strength of rVIII-SingleChain after 3 to 6 months. Subjects from Parts 2 and 3 participating in the surgical substudy received an individualized dose regimen of rVIII-SingleChain, based on the type of surgery and the clinical status of the subject.
  Other Names: Recombinant Factor VIII (rFVIII); CSL627
Biological: Octocog alfa — In Part 1 of the study, subjects received a single intravenous infusion of 50 IU/kg of octocog alfa preceded by a 4-day washout period. Octocog alfa is the international nonproprietary name (INN) for recombinant human coagulation factor VIII.
  Other Names: Human coagulation factor VIII (rDNA)

SUMMARY:
This is an open-label, non-randomized, efficacy, safety and pharmacokinetic (PK) study comparing octocog alfa and rVIII-SingleChain. The study consists of three parts, a PK period (Part 1), a continuation of dosing safety and efficacy period (Part 2) and a safety, efficacy, and repeat PK period (Part 3) and also includes a surgical sub-study for subjects enrolled in Parts 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe hemophilia A defined as <1% FVIII:C documented in medical records.
* Males between 18 and 65 years of age (Parts 1 and 2).
* Males between 12 and 65 years of age (Part 3).
* Subjects who have received or are currently receiving FVIII products (plasma-derived and/or recombinant FVIII) and have had >150 exposure days (EDs) with a FVIII product
* Written informed consent for study participation obtained before undergoing any study specific procedures.

Exclusion Criteria:

* Any history of or current FVIII inhibitors
* Any first order family history of FVIII inhibitors
* Use of an Investigational Medicinal Product within 30 days prior to the first rVIII-SingleChain administration.
* Administration of any cryoprecipitate, whole blood or plasma within 30 days prior to administration of rVIII-SingleChain or reference product.
* Known hypersensitivity (allergic reaction or anaphylaxis) to any FVIII product or hamster protein.
* Any known congenital or acquired coagulation disorder other than congenital FVIII deficiency.
* Platelet count < 100,000/µL at screening.
* Human immunodeficiency virus (HIV) positive subjects with a CD4 count < 200/mm3, in their medical history or at screening if available results are older than one year. (HIV positive subjects may participate in the study and antiviral therapy are permitted, at the discretion of the Investigator).
* Subject currently receiving IV immunomodulating agents such as immunoglobulin or chronic systemic corticosteroid treatment.
* Subject with serum aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT) values > 5 times (x) the upper limit of normal (ULN) at Screening.
* Subjects with serum creatinine values > 2 x ULN at Screening.
* Evidence of thrombosis, including deep vein thrombosis, stroke, pulmonary embolism, myocardial infarction and arterial embolus within 3 months prior to Day 1.
* Experienced life-threatening bleeding episode or had major surgery or an orthopedic surgical procedure during the 3 months prior to Day 1.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (54):
- United States (9):
  - Study Site, Sacramento, California
  - Study Site, San Diego, California
  - Study Site, Aurora, Colorado
  - Study Site, Hartford, Connecticut
  - Study Site, Miami, Florida
  - Study Site, Chicago, Illinois
  - Study Site, New Orleans, Louisiana
  - Study Site, Houston, Texas
  - Study Site, Milwaukee, Wisconsin
- Australia (2):
  - Study Site, Nedlands
  - Study Site, Perth
- Austria (2):
  - Study Site, Graz
  - Study Site, Vienna
- Study Site, New Brunswick, Canada
- Study Site, Hradec Králové, Czechia
- Germany (6):
  - Study Site, Berlin
  - Study Site, Bonn
  - Study Site, Giessen
  - Study Site, Hamburg
  - Study Site, Hanover
  - Study Site, Heidelberg
- Study Site, Debrecen, Hungary
- Italy (4):
  - Study Site, Florence
  - Study Site, Milan
  - Study Site, Padua
  - Study Site, Torino
- Japan (8):
  - Study Site, Kashihara, Nara
  - Study Site, Kitakyushu, Fukuoka
  - Study Site, Nagoya
  - Study Site, Nishinomiya, Hyogo
  - Study Site, Okayama
  - Study Site, Saitama
  - Study Site, Suginami-ku, Tokyo
  - Study Site, Tokyo
- Study Site, Beirut, Lebanon
- Study Site, Kuala Lumpur, Malaysia
- Study Site, Utrecht, Netherlands
- Philippines (2):
  - Study Site, Cebu City
  - Study Site, Davao City
- Poland (3):
  - Study Site, Wroclaw, Silesian Voivodeship
  - Study Site, Gdansk
  - Study Site, Krakow
- Study Site, Bucharest, Romania
- Russia (2):
  - Study Site, Barnaul
  - Study Site, Kemerovo
- South Africa (2):
  - Study Site, Cape Town
  - Study Site, Johannesburg
- Spain (3):
  - Study Site, A Coruña
  - Study Site, Barcelona
  - Study Site, Valencia
- Ukraine (3):
  - Study Site, Dnipropetrovsk
  - Study Site, Donetsk
  - Study Site, Lviv
- Study Site, London, United Kingdom

REFERENCES:
- [Derived] Mahlangu J, Kuliczkowski K, Karim FA, Stasyshyn O, Kosinova MV, Lepatan LM, Skotnicki A, Boggio LN, Klamroth R, Oldenburg J, Hellmann A, Santagostino E, Baker RI, Fischer K, Gill JC, P'Ng S, Chowdary P, Escobar MA, Khayat CD, Rusen L, Bensen-Kennedy D, Blackman N, Limsakun T, Veldman A, St Ledger K, Pabinger I; AFFINITY Investigators. Efficacy and safety of rVIII-SingleChain: results of a phase 1/3 multicenter clinical trial in severe hemophilia A. Blood. 2016 Aug 4;128(5):630-7. doi: 10.1182/blood-2016-01-687434. Epub 2016 Jun 21. PMID 27330001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, multinational study enrolled subjects at 54 participating study centers in the United States, Japan, Europe, Australia, Canada, Lebanon, Malaysia, Philippines, Russian Federation, South Africa, and Ukraine.
Pre-assignment Details: Screening took place 4 to 28 days prior to first dose of study product (rVIII-SingleChain). A total of 204 subjects were screened, 29 of these did not fulfill all eligibility criteria and were therefore screening failures. A total of 175 subjects were enrolled; 174 subjects were exposed to treatment with rVIII-SingleChain.
Groups:
- Recombinant Factor VIII (rFVIII): In Part 1 of the study (a single-sequence crossover pharmacokinetic [PK] analysis), 27 subjects received a single injection of octocog alfa followed by a single injection of rVIII-SingleChain. Twenty-six of the 27 subjects from Part 1 then entered Part 2 of the study where they were assigned either to an on-demand or prophylaxis regimen with repeat injections of rVIII-SingleChain until they reached 50 exposure days (EDs). In Part 3 of the study, 148 additional subjects were enrolled and were assigned either to an on-demand or prophylaxis regimen with repeat injections of rVIII-SingleChain until they reached 50 EDs; 64 of these subjects participated in additional PK analyses. Overall, 174 subjects received rVIII-SingleChain as either on-demand or prophylaxis regimens, and 13 subjects participated in the surgical substudy.
Period: Overall Study
Arm/Group | Recombinant Factor VIII (rFVIII)
Started | 174
Completed | 161
Not Completed | 13
Not completed — Knee surgery (prior to surgery substudy) | 1
Not completed — Physician Decision | 1
Not completed — 50 Exposure days not reached | 2
Not completed — Withdrawal by Subject | 8
Not completed — Subject did not reach 6 mo of treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- Recombinant Factor VIII (rFVIII): In Part 1 of the study (a single-sequence crossover PK analysis), 27 subjects received a single injection of octocog alfa followed by a single injection of rVIII-SingleChain. Twenty-six of the 27 subjects from Part 1 then entered Part 2 of the study where they were assigned either to an on-demand or prophylaxis regimen with repeat injections of rVIII-SingleChain until they reached 50 EDs. In Part 3 of the study, 148 additional subjects were enrolled and were assigned either to an on-demand or prophylaxis regimen with repeat injections of rVIII-SingleChain until they reached 50 EDs; 64 of these subjects participated in additional PK analyses. Overall, 174 subjects received rVIII-SingleChain as either on-demand or prophylaxis regimens, and 13 subjects participated in the surgical substudy.
Arm/Group | Recombinant Factor VIII (rFVIII)
Number analyzed (Participants) | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (11.77)
Age, Customized [Number; unit: participants]
  Adolescents (12-17 years) | 14
  Adults (18-65 years) | 160
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 174
Type of FVIII product used before enrollment [Number; unit: participants] — Type of FVIII product used by the subjects before enrollment into the study. This could have been a plasma-derived FVIII product or a recombinant FVIII product.
  participants
    Plasma-derived Product | 83
    Recombinant Product | 91
Treatment modality of FVIII therapy before enrollment [Number; unit: participants] — Treatment modality of FVIII therapy before enrollment, ie, routine prophylaxis or on-demand treatment. If a subject used both modalities, only the most recent one was counted.
  participants
    Prophylaxis | 82
    On-demand | 92

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success
Description: The investigator rated the efficacy of the treatment based on a 4-point rating scale "excellent, good, moderate or poor/no response". Efficacy ratings of "excellent" or "good" were considered treatment success for this end point; the percentage of bleeding events with a rating of excellent or good and the 95% confidence interval are presented. The denominator includes all treated bleeding events. The 95% confidence interval is based on a model to account for within-subject correlation.
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: % bleeding events successfully treated
Units Other Than Participants: Number of treated bleeding events
Groups:
- rVIII-SingleChain On-demand: The rVIII-SingleChain On-demand group consisted of all subjects in the efficacy population who received at least 1 dose rVIII-SingleChain as part of on-demand treatment during Parts 2 or 3 of the study. There were 27 subjects in the rVIII-SingleChain On-demand group.
- rVIII-SingleChain Prophylaxis: The rVIII-SingleChain Prophylaxis group consisted of all subjects in the efficacy population who received at least 1 dose rVIII-SingleChain as part of routine prophylaxis treatment during Parts 2 or 3 of the study. There were 146 subjects in the rVIII-SingleChain Prophylaxis group.
- rVIII-SingleChain: The Efficacy population consisted of all subjects who received at least 1 dose of rVIII-SingleChain as part of either routine prophylaxis treatment or on-demand treatment during Parts 2 or 3 of the study. There were 173 subjects in the Efficacy population.
Arm/Group | rVIII-SingleChain On-demand | rVIII-SingleChain Prophylaxis | rVIII-SingleChain
Number analyzed (Participants) | 27 | 146 | 173
Number analyzed (Number of treated bleeding events) | 590 | 258 | 848
% bleeding events successfully treated | 92.4 [87.8 to 95.3] | 92.2 [86.3 to 95.8] | 92.3 [88.9 to 94.8]

2. Primary Outcome: Inhibitor Formation to FVIII
Description: Number of subjects who develop inhibitors to FVIII
Time Frame: Up to 24 months
Measure: Number; unit: participants
Arm/Group | Recombinant Factor VIII (rFVIII)
Number analyzed (Participants) | 174
participants | 0

3. Primary Outcome: Annualized Spontaneous Bleeding Rate
Description: The annualized spontaneous bleeding rate (AsBR) was derived for each subject as follows: 365.25*(number of spontaneous bleeding episodes requiring treatment) / (observed treatment period of interest).
Time Frame: Up to 24 months
Measure: Median (Inter-Quartile Range); unit: Number of spontaneous bleeds per year
Arm/Group | rVIII-SingleChain On-demand | rVIII-SingleChain Prophylaxis
Number analyzed (Participants) | 27 | 146
Number of spontaneous bleeds per year | 11.73 [2.8 to 36.5] | 0.00 [0.0 to 2.4]
Statistical Analysis 1: Comparison: rVIII-SingleChain On-demand vs rVIII-SingleChain Prophylaxis; A test of the null hypothesis of no difference on AsBR between the 2 comparison groups was based on the Poisson Regression method. The corresponding prophylaxis/on-demand ratio with 95% confidence interval (CI) was calculated; Test type: Superiority or Other; p < 0.0001, Poisson, regression; Rate ratio = 0.08, 95% CI 2-sided [0.07 to 0.10]

4. Primary Outcome: Treatment Success During the Peri-operative Surgical Sub-study
Description: Subjects received rVIII-SingleChain before and during surgery based on the type of surgery and the clinical status of the subject. The investigator rated the efficacy of the treatment based on a 4-point surgical treatment rating scale of "excellent, good, moderate or poor/no response". Efficacy ratings of "excellent" or "good" were considered treatment success for this end point. The rate of success, defined as the percentage of surgeries with a rating of excellent or good for hemostatic efficacy on the surgical treatment scale is presented for the Surgical Population, based on the total number of surgeries (N=16) as denominator.
Time Frame: From the start of surgery through the post-operative recovery (generally up to 14 days after surgery)
Measure: Number; unit: % of surgeries with successful treatment
Groups:
- rVIII-SingleChain Surgical: The rVIII-SingleChain Surgical group included all subjects enrolled in the surgical sub-study who received at least 1 dose of rVIII-SingleChain during the surgical sub-study. There were 13 subjects in the rVIII-SingleChain Surgical group.
Arm/Group | rVIII-SingleChain Surgical
Number analyzed (Participants) | 13
% of surgeries with successful treatment | 100

5. Secondary Outcome: AUC0-∞ (Part 1)
Description: AUC0-∞ (AUC from 0 extrapolated to infinity) of a single infusion of octocog alfa and rVIII-SingleChain without correction for subject's predose plasma FVIII activity. FVIII activity values for octocog alfa are dose-adjusted for chromogenic potency.
Time Frame: Before infusion and at up to 10 time points within 72 hours of infusion
Measure: Mean (Standard Deviation); unit: IU*h/dL
Groups:
- PK Population (Part 1): The PK population (Part 1) consisted of subjects who had received 1 dose of 50 IU/kg of rVIII-SingleChain and for whom a sufficient number of analyzable PK samples were obtained to permit the evaluation of the PK profile. In the Part 1 PK analysis, these subjects also received 1 dose of 50 IU/kg octocog alfa. There were 27 subjects in the PK population (Part 1).
Arm/Group | PK Population (Part 1)
Number analyzed (Participants) | 27
IU*h/dL
  Octocog alfa | 1550 (552)
  rVIII-SingleChain | 2090 (650)

6. Secondary Outcome: Cmax (Part 1)
Description: Cmax of a single infusion of octocog alfa and rVIII-SingleChain with correction for subject's predose plasma FVIII activity. FVIII activity values for octocog alfa are dose-adjusted for chromogenic potency.
Time Frame: Before infusion and at up to 10 time points within 72 hours of infusion
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | PK Population (Part 1)
Number analyzed (Participants) | 27
IU/dL
  Octocog alfa | 116 (18.1)
  rVIII-SingleChain | 113 (17.4)

7. Secondary Outcome: Tmax (Part 1)
Description: Tmax = time of Cmax (with correction for subject's predose plasma FVIII activity) after a single infusion of octocog alfa and rVIII-SingleChain.
Time Frame: Before infusion and at up to 10 time points within 72 hours of infusion
Measure: Median (Full Range); unit: hours
Arm/Group | PK Population (Part 1)
Number analyzed (Participants) | 27
hours
  Octocog alfa | 0.583 [0.450 to 0.800]
  rVIII-SingleChain | 0.683 [0.467 to 1.25]

8. Secondary Outcome: Half-life (t1/2) (Part 1)
Description: Half-life (t1/2) of a single infusion of octocog alfa and rVIII-SingleChain without correction for subject's predose plasma FVIII activity.
Time Frame: Before infusion and at up to 10 time points within 72 hours of infusion.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PK Population (Part 1)
Number analyzed (Participants) | 27
hours
  Octocog alfa | 13.3 (4.36)
  rVIII-SingleChain | 14.5 (3.77)

9. Secondary Outcome: Mean Residence Time (MRT) (Part 1)
Description: Mean residence time (MRT) of a single infusion of octocog alfa and rVIII-SingleChain without correction for subject's predose plasma FVIII activity.
Time Frame: Before infusion and at up to 10 time points within 72 hours of infusion
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PK Population (Part 1)
Number analyzed (Participants) | 27
hours
  Octocog alfa | 17.1 (5.57)
  rVIII-SingleChain | 20.4 (5.49)

10. Secondary Outcome: Clearance (Cl) (Part 1)
Description: Clearance (Cl) of a single infusion of octocog alfa and rVIII-SingleChain without correction for subject's predose plasma FVIII activity. FVIII activity values for octocog alfa are dose-adjusted for chromogenic potency.
Time Frame: Before infusion and at up to 10 time points within 72 hours of infusion
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | PK Population (Part 1)
Number analyzed (Participants) | 27
mL/h/kg
  Octocog alfa | 3.68 (1.41)
  rVIII-SingleChain | 2.64 (0.846)

11. Secondary Outcome: Volume of Distribution at Steady-state (Vss) (Part 1)
Description: Volume of distribution at steady-state (Vss) of a single infusion of octocog alfa and rVIII-SingleChain without correction for subject's predose plasma FVIII activity. FVIII activity values for octocog alfa are dose-adjusted for chromogenic potency.
Time Frame: Before infusion and at up to 10 time points within 72 hours of infusion
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | PK Population (Part 1)
Number analyzed (Participants) | 27
mL/kg
  Octocog alfa | 57.1 (11.3)
  rVIII-SingleChain | 50.0 (7.51)

12. Secondary Outcome: Incremental Recovery (Part 1)
Description: Incremental recovery of a single infusion of octocog alfa and rVIII-SingleChain with correction for subject's predose plasma FVIII activity. FVIII activity values for octocog alfa are dose-adjusted for chromogenic potency.
Time Frame: At 30 minutes after infusion
Measure: Mean (Standard Deviation); unit: [IU/dL]/[IU/kg]
Arm/Group | PK Population (Part 1)
Number analyzed (Participants) | 27
[IU/dL]/[IU/kg]
  Octocog alfa | 2.32 (0.381)
  rVIII-SingleChain | 2.24 (0.357)

13. Secondary Outcome: Annualized Bleeding Rate for Total Bleeds and Traumatic Bleeds
Description: The annualized bleeding rate was derived for each subject as follows: 365.25*(number of bleeding episodes requiring treatment) / (observed treatment period of interest).
Time Frame: Up to 24 months
Measure: Median (Inter-Quartile Range); unit: Number of bleeds per year
Arm/Group | rVIII-SingleChain On-demand | rVIII-SingleChain Prophylaxis
Number analyzed (Participants) | 27 | 146
Number of bleeds per year
  Total Bleeds | 19.64 [6.2 to 46.5] | 1.14 [0.0 to 4.2]
  Traumatic Bleeds | 3.12 [0.0 to 8.4] | 0.00 [0.0 to 0.9]

14. Secondary Outcome: Proportion of Bleeding Episodes Requiring 1, 2, 3 or > 3 Infusions of rVIII-SingleChain to Achieve Hemostasis
Description: Percentage of bleeding episodes requiring 1, 2, 3 or > 3 infusions of rVIII-SingleChain to achieve hemostasis. The denominator includes all treated bleeding episodes.
Time Frame: During the study (up to 24 months; assessed at Months 1, 2, 3, 4, 5, 6, 9, 12, 15, 18, 21 and 24)
Measure: Number; unit: Percentage of bleeding episodes
Units Other Than Participants: Treated bleeding episodes
Groups:
- rVIII-SingleChain: The Efficacy population consisted of all subjects who received at least one dose of rVIII-SingleChain as part of either routine prophylaxis treatment or on-demand treatment during Parts 2 or 3 of the study. There were 173 subjects in the Efficacy population.
Arm/Group | rVIII-SingleChain On-demand | rVIII-SingleChain Prophylaxis | rVIII-SingleChain
Number analyzed (Participants) | 27 | 146 | 173
Number analyzed (Treated bleeding episodes) | 590 | 258 | 848
Percentage of bleeding episodes
  Requiring 1 infusion for hemostasis | 82.7 | 76.7 | 80.9
  Requiring 2 infusions for hemostasis | 12.0 | 14.0 | 12.6
  Requiring 3 infusions for hemostasis | 3.22 | 3.88 | 3.42
  Requiring >3 infusions for hemostasis | 2.03 | 5.43 | 3.07

15. Other Pre Specified Outcome: Incremental Recovery (Part 3)
Description: Incremental recovery of an initial and repeat infusion of rVIII-SingleChain with correction for subject's predose plasma FVIII activity.
Time Frame: At 30 minutes after infusion
Measure: Mean (Standard Deviation); unit: [IU/dL]/[IU/kg]
Groups:
- rVIII-SingleChain PK Population (Part 3): The rVIII-SingleChain PK population (Part 3) consisted of subjects who received rVIII-SingleChain during Part 3 of the study (initial and repeat dose) and for whom a sufficient number of analyzable PK samples were obtained to permit the evaluation of the PK profile. In Part 3, 64 subjects participated in the initial PK, of whom 30 also participated in the repeat PK.
Arm/Group | rVIII-SingleChain PK Population (Part 3)
Number analyzed (Participants) | 63
[IU/dL]/[IU/kg]
  Initial, n = 63 | 1.85 (0.404)
  Repeat, n = 29 | 1.99 (0.352)

16. Other Pre Specified Outcome: Volume of Distribution at Steady-state (Vss) (Part 3)
Description: Volume of distribution at steady-state (Vss) of an initial and repeat infusion of rVIII-SingleChain without correction for subject's predose plasma FVIII activity.
Time Frame: Before infusion and at up to 12 time points within 96 hours of infusion.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | rVIII-SingleChain PK Population (Part 3)
Number analyzed (Participants) | 64
mL/kg
  Initial, n = 64 | 59.5 (14.2)
  Repeat, n = 30 | 53.1 (8.74)

17. Other Pre Specified Outcome: Clearance (Cl) (Part 3)
Description: Clearance (Cl) of an initial and repeat infusion of rVIII-SingleChain without correction for subject's predose plasma FVIII activity.
Time Frame: Before infusion and at up to 12 time points within 96 hours of infusion.
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | rVIII-SingleChain PK Population (Part 3)
Number analyzed (Participants) | 64
mL/h/kg
  Initial, n = 64 | 3.15 (1.21)
  Repeat, n = 30 | 3.05 (1.1)

18. Other Pre Specified Outcome: Mean Residence Time (MRT) (Part 3)
Description: Mean residence time (MRT) of an initial and repeat infusion of rVIII-SingleChain without correction for subject's predose plasma FVIII activity.
Time Frame: Before infusion and at up to 12 time points within 96 hours of infusion.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | rVIII-SingleChain PK Population (Part 3)
Number analyzed (Participants) | 64
hours
  Initial, n = 64 | 20.3 (5.36)
  Repeat, n = 30 | 18.9 (5.39)

19. Other Pre Specified Outcome: Half-life (t1/2) (Part 3)
Description: Half-life (t1/2) of an initial and repeat infusion of rVIII-SingleChain without correction for subject's predose plasma FVIII activity.
Time Frame: Before infusion and at up to 12 time points within 96 hours of infusion.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | rVIII-SingleChain PK Population (Part 3)
Number analyzed (Participants) | 64
hours
  Initial, n = 64 | 14.1 (3.82)
  Repeat, n = 30 | 12.9 (3.7)

20. Other Pre Specified Outcome: Tmax (Part 3)
Description: Tmax = time of Cmax (with correction for subject's predose plasma FVIII activity) after an initial and repeat infusion of rVIII-SingleChain.
Time Frame: Before infusion and at up to 12 time points within 96 hours of infusion.
Measure: Median (Full Range); unit: hours
Arm/Group | rVIII-SingleChain PK Population (Part 3)
Number analyzed (Participants) | 63
hours
  Initial, n = 63 | 0.333 [0.117 to 1.22]
  Repeat, n = 29 | 0.317 [0.117 to 0.667]

21. Other Pre Specified Outcome: Cmax (Part 3)
Description: Cmax of an initial and repeat infusion of rVIII-SingleChain with correction for subject's predose plasma FVIII activity.
Time Frame: Before infusion and at up to 12 time points within 96 hours of infusion
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | rVIII-SingleChain PK Population (Part 3)
Number analyzed (Participants) | 63
IU/dL
  Initial, n = 63 | 99.9 (19.9)
  Repeat, n = 29 | 108 (18.5)

22. Other Pre Specified Outcome: AUC0-∞ (Part 3)
Description: AUC0-∞ (AUC from 0 extrapolated to infinity) of an initial and repeat infusion of rVIII-SingleChain without correction for subject's predose plasma FVIII activity.
Time Frame: Before infusion and at up to 12 time points within 96 hours of infusion
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | rVIII-SingleChain PK Population (Part 3)
Number analyzed (Participants) | 64
IU*h/dL
  Initial, n = 64 | 1830 (640)
  Repeat, n = 30 | 1880 (649)

ADVERSE EVENTS:
Time Frame: For the duration of the study, approximately 2 years, 10 months.
Description: The Safety Population comprised all subjects treated with rVIII-SingleChain. A total of 14592 rVIII-SingleChain infusions were administered to 174 subjects during the study.
Groups:
- Safety Population: The Safety Population comprised all subjects treated with rVIII-SingleChain.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 8/174
Other Adverse Events (participants affected / at risk) | 45/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=174)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=174)
Headache (Nervous system disorders) | 13 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (22)
Nasopharyngitis (Infections and infestations) | 18 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.